CLINICAL TRIAL: NCT00059709
Title: Understanding and Learning How to Resolve Family Conflict
Brief Title: Learning to Resolve Family Conflict
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 5R01HD38895-2; 5R01HD038895 (NIH)
Record Dates: First submitted 2003-05-02; First posted 2003-05-05 (Estimated); Last update posted 2007-04-03 (Estimated); Status verified 2006-01

CONDITIONS: Conflict; Family Relations
Keywords: Conflict Resolution training; Children

INTERVENTIONS:
Procedure: Mediated Negotiation Training

SUMMARY:
This study will evaluate the effectiveness of conflict resolution training for families with preschool and elementary school-aged children.

DETAILED DESCRIPTION:
This study will examine the language, reasoning, and social skills used by preschool and elementary school children when they and their parents attempt to understand, conduct, and resolve disputes in everyday family interaction. Families will be given conflict resolution training designed to promote listening and speaking skills that result in more accurate interpersonal and emotional understanding. The training may lower the emotional volatility of family interaction, lower the rate of arguing and fighting between parents and children, increase the rate and frequency of verbal negotiation, and encourage the adoption of conflict strategies that focus on future-oriented behavior and positive outcomes.

A total of 324 working class families, representative of the primary ethnic populations in Chicago (African American, Caucasian, and Mexican American), will be selected for participation. Both parents, one 4- to 6-year-old child, and one 6- to 8-year-old sibling will participate. Single parent families will also be included; the parent will be asked to nominate a second adult or an additional older sibling in place of the second parent.

Each family proceeds through three phases. The initial phase allows assessment of conflict histories, good times, self-appraisals of psychological well-being, affective and social variables that operate within the family, and the family members' ability to discuss and negotiate ongoing problems.

In the second phase, families are randomly assigned to one of three experimental conditions. One group is given conflict resolution training and then participates in a series of tasks that focus on child-parent narration, negotiation, and negotiation assessments. A second group participates in the same tasks without training. A third group undergoes only the negotiation assessments. The effectiveness of the training will be evaluated by experimentally assessing conflict resolution skills before and after training in both home and school contexts.

The third phase is a six-month follow-up visit, during which parents and children are again observed negotiating problems. Psychological well-being and affective feelings are once again assessed. The study ends with a debriefing interview for the parents.

The study consists of 14 study visits. Each member in the family will also have four training sessions. Visits are scheduled 3 to 4 times a month, depending on the family's availability.

ELIGIBILITY:
Inclusion Criteria:

* Nuclear family with at least one biological parent
* African American, Caucasian, or Mexican American
* At least two children: one between the ages of 4 and 6 years, and one between the ages of 6 and 10 years

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Stein, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States